CLINICAL TRIAL: NCT06269250
Title: Acceptance and Perceived Benefits of Digitalization by Medical Assistants (ANDI-MFA)
Brief Title: Acceptance and Perceived Benefits of Digitalization by Medical Assistants
Acronym: ANDI-MFA
Status: Recruiting | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Mirjam Jansen; medmedia Academy (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANDI-MFA2023_10
Record Dates: First submitted 2023-10-22; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Health Care Providers; Patient Safety; eHealth
Keywords: digital processes; e-prescriptions; health care providers; medical assistants; acceptance; life-long learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sample assessed in Wave 2023: Participants can be any healthcare worker, including dental and medical assistants, aged 18 or older.
  Interventions: Other: Policy Change
- sample assessed in Wave 2024: Participants can be any healthcare worker, including dental and medical assistants, aged 18 or older.
  Interventions: Other: Policy Change

INTERVENTIONS:
Other: Policy Change — There will be a change with the digitalization in the health care system with the beginning of the year 2024 and between Wave 1 and Wave 2

SUMMARY:
The aim of this project is to improve the integration of digital processes, including e-prescriptions, within medical and dental practices for healthcare professionals. Through a better understanding of the obstacles healthcare workers encounter during the adoption of digital processes and their feedback post-implementation, this study will add to the current state of science, contributing to digital process optimization in healthcare.

DETAILED DESCRIPTION:
This study uses an online questionnaire to collect data from respondents regarding their experiences and observations as healthcare professionals in the implementation of digital processes, as well as their perception of digital processes post-implementation. The survey will be conducted at two different time points, in 2023 and 2024. As part of this initiative, we plan to share the feedback and recommendations gathered with the Federal Minister of Health and relevant authorities in collaboration with GEMATIK.

Main research questions are

I. What challenges do healthcare professionals encounter in the implementation of digital processes? II. How can the offers for the implementation and introduction of digital processes (e.g. e-prescription) in medical practice for medical and dental professionals be supported and optimized? III. What changes from the first measurement wave in 2023 to the second in 2024 with regard to the perception of digital offers, experiences, and observations?

ELIGIBILITY:
Inclusion Criteria:

- Ability to participate in surveys (e.g., sufficient German or English language skills)

Exclusion Criteria:

* Younger than 18 years
* Illiteracy
* Massively limited cognitive abilities, i.e., linguistic components of the digital offerings must be able to be used to complete questionnaires or participate in interviews

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Health Care Workers, including medical assistances
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adoption and acceptance of information technology (IT) | 3 months
  The items assess the adoption and acceptance of telematic infrastructure (TI) in medical or dental practices. They collect data on the use of TI, its impact on daily operations, and its acceptance. These are example items for each category:
  1. Is your medical office connected to the Telematics Infrastructure (TI)? (Answer options: "bot at all", "some days", "more than half of the days", "almost every day")
  2. Does the TI connection run smoothly without causing disruption to your practice operations? (Answer options: "not at all", "some days", "more than half of the days", "almost every day")
  3. Do you know if your (dental) office management fundamentally rejects a TI connection? (Answer options: "I strongly disagree", "I disagree", "I agree", "I strongly agree", "I don't know")
Requests by patients regarding IT | 3 months
  The items assess the frequency of patients' inquiries about various digital health applications and services. These are example items:
  1. How often have been asked by patients about an e-prescription? (Answer options: "not at all", "some days", "more than half of the days", "almost every day")
  2. What topics are you most frequently asked about by your patients? (Answer options: "online medical consultation", "eAU", "e-prescription", "ePA", "digital health apps (DIGAs)", "fitness trackers like smartwatches")
Perceived Benefits of IT | 3 months
  The perceived benefits of IT are measured through self-report

SECONDARY OUTCOMES:
Knowledge and Digital health literacy | 3 months
  The items assess the participants' awareness and knowledge of digital health tools and their ability to access and comprehend health-related information. Example items are:
  1. Have you heard of TI applications such as eAU, KIM, e-prescription, ePA, etc.? (Answer options: "I strongly disagree", "I disagree", "I agree", "I strongly agree", "I don't know")
  2. Have you heard of "ePA for all"? (Answer options: "I strongly disagree", "I disagree", "I agree", "I strongly agree", "I don't know.") If yes, do you feel well-informed enough to answer questions from patients about it? If no, do you know the informational materials for the waiting room or from another source such as gematik, e.g., regarding e-prescription?
  3. Do you know the three redemption methods for the e-prescription? (Answer options: "I strongly disagree", "I disagree", "I agree", "I strongly agree", "I don't know")
Preferred learning format | 3 months
  The items assess how healthcare professionals prefer to access information related to their work and digital health applications. Example items are:
  1. How often do you actively search the internet for information about digital applications? (Answer options: "never", "almost never", "sometimes", "almost daily", "daily")
  2. On which platforms do you seek information when looking for details about digital health applications? (Answer options: Facebook, Facebook group, LinkedIn, Instagram, TikTok, Xing, other)
  3. How do you prefer to inform yourself about applications related to your work? (multiple answer option)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Dahmen, Dr. med., Study Director — Constructor University Bremen gGmbH
Locations (1):
- Germany, Bremen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project Partner — http://medmedia.koeln
- See also: Main PI — https://constructor.university/sonia-lippke